CLINICAL TRIAL: NCT04204824
Title: The Effectiveness of Ultrasound Treatment in the Management of Plantar Fasciitis: A Randomized, Placebo-Controlled Study
Brief Title: Ultrasound Treatment in the Management of Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Sage Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 399-2015-2016
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — High-Energy Shock Waves; Exercise

STUDY DESIGN:
Intervention Model Description: Two groups: Control vs. experimental
Who Masked: Participant, Investigator
Masking Description: An independent investigator will set the parameters with the machine outside the treatment area and not in sight of the principal investigator or participant. The face of the machine will then be covered so neither the principal investigator nor the participant can see the settings.The principal investigator and the participants will not be aware of their group assignments until conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound and exercise (Experimental): This group will receive ultrasound treatment, strengthening exercises and stretching exercises.
  Interventions: Other: Ultrasound and exercise
- Sham Ultrasound and exercise (Active Comparator): This group will receive sham ultrasound treatment, strengthening exercises and stretching exercises.
  Interventions: Other: Ultrasound and exercise

INTERVENTIONS:
Other: Ultrasound and exercise — The control group's ultrasound will be set at an intensity of 0 w/cm2. The first 3 treatments to the experimental group will be continuous ultrasound with an intensity of 1.0w/cm2 for 7 minutes. The next 6 treatments for the experimental group (2 times a week for 3 weeks) will have pulsed ultrasound at an intensity of 1.0w/cm2 with a 50% (1:1) duty cycle for 10 minutes. All will have a frequency of 3 MHZ.
  All participants in each group will be given specific exercises targeting intrinsic and extrinsic muscles of the foot and ankle. Exercises will be performed with a level of thera-band that is challenging to the individual participant in each plane of motion without increased pain for 3 sets of 10 repetitions each and one time each day independently at home during the duration of the treatment protocol (4 weeks) and recorded in an exercise log diary Specific stretches for the plantar fascia and Achilles tendon will be performed 3 times each for 30 second intervals and at home

SUMMARY:
The purpose of this study is to examine the effectiveness of ultrasound treatment in addition to an exercise program to improve pain and function in individuals with plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is a common cause of foot pain, affecting an estimated 2 million people per year.1 Although there are large numbers of people seeking medical attention for this condition, there remains some confusion among health care providers as to the most efficacious treatment and some authors conclude that no data solidly supports effectiveness of treatment.2 Few randomized control studies have been published with respect to treatment of PF with ultrasound. Only one study of this nature was published in 1995 by Crawford et al.3 This research found the true ultrasound was no more effective then sham ultrasound and the authors concluded that future studies need to clarify ultrasound parameters with respect to intensity, duty cycle, frequency, area, duration, dosage, and treatment size.

The purpose of this study is to examine the effectiveness of ultrasound treatment in addition to an exercise program to improve pain and function in individuals with plantar fasciitis. The investigator's primary hypothesis is individuals with PF will show a greater improvement in pain and function with ultrasound and an exercise program as compared to just an exercise program alone.

Research Questions for each outcome measure:

1. Following the four week intervention period, the experimental or the True Ultrasound group (TUG) group will show a greater improvement in their pain rating during two different time intervals: Pain in the previous 24 hours and with initial steps in the morning, as well as three different functional activities: Pain during single limb stance, 30 minutes of standing during ADLs, and walking 1000meter (.62miles) according to the Visual Analog Scale (VAS) compared to the control group.

2 Following the four week intervention period, the experimental group, TUG, will show an improved percentage of level of function in ADLs and sports as measured by the Foot and Ankle Ability Measure (FAAM) as compared to the control group.

3 Following the four week intervention period the experimental group, TUG, will demonstrate an improved range of motion (ROM) of ankle dorsiflexion in subtalar neutral as measured by a goniometer as compared to the control group.

4 Following a four week intervention period the experimental group, TUG, will demonstrate an increase in ankle strength of the Anterior Tibialis, Posterior Tibialis, Peroneus Longus, Peroneus Brevis, and Gastrocnemius as measured by a hand held dynamometer as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* a progressive onset of heel pain lasting 6 months or less, localized to the medial calcaneal tubercle and pain with first steps in the morning.

Exclusion Criteria:

* all patients currently receiving treatment for plantar fasciitis within the last 6 months including night splints, orthotic management, iontophoresis with dexamethasone or acetic acid, corticosteroid injections, extracorporeal shock wave laser therapy, microwave diathermy, radiotherapy, stereotactic radiofrequency, trigger-point needling with infiltration, and ultrasound.
* Participants with numbness or tingling with or without provocation in the lower extremity, undiagnosed pain, strength impairment of the ankle of less than a 3+/5 measured with specific manual muscle tests
* pregnant women
* Participants with Type I or II Diabetes Mellitis, systemic inflammatory arthritis, cancer, active tuberculosis, psoriasis, decreased circulation, infections, cemented joint replacements
* patients with pacemakers, thrombophlebitis, uncontrolled bleeding or taking blood thinning medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale for pain | Change measures (baseline and up to 5 weeks)
  The Visual Analog Scale will be used to measure pain at the initial evaluation and at the conclusion of the study for the following intervals: 1) over the previous 24 hour period, 2) with the initial steps first thing in the morning, 3) in single limb stance, 4) after standing for 30 minutes in the course of the participants normal standing activities, and 5) after walking for 1000 meters. This scale has a minimum value of 0 and a maximum value of 10. Higher scores mean worst outcomes.
Function | Change measures (baseline and up to 5 weeks)
  The Foot and Ankle Ability Measure is a functional outcome measure validated in the physical therapy setting.7 It will be used to measure differences in ability in activities of daily living and sports at the initial evaluation and at the conclusion of the study. The final score is reported in % (100% being the maximum value). Higher scores reflect better outcomes.
Strength | Change measures (baseline and up to 5 weeks)
  Strength will be measured with a hand held dynamometer for the tibialis anterior, tibialis posterior, peroneus longus and brevis, and gastrocnemius.
Range of Motion | Change measures (baseline and up to 5 weeks)
  Dorsiflexion active range of motion (AROM) and dorsiflexion passive range of motion (PROM) measurements will be collected at the initial evaluation and at the conclusion of the treatment protocol. Dorsiflexion AROM and PROM will be measured in prone with the forefoot aligned in the frontal plane, the subtalar joint in neutral, the goniometer measuring the sagittal plane with the proximal arm aligned with the fibular head and the distal arm aligned along the lateral border of the 5th metatarsal by the principal investigator.

IPD SHARING:
Plan to Share IPD: No